CLINICAL TRIAL: NCT01500876
Title: A Feasibility Study Using Four-Dimensional CT Imaging to Evaluate Lung Strain in Patients Treated With External Beam Radiation Therapy for Primary Lung Cancer
Brief Title: A Feasibility Study Using Four-Dimensional CT Imaging for Primary Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Neal Edward Dunlap, Associate Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCC-RAD-11-02
Record Dates: First submitted 2011-12-05; First posted 2011-12-29 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Lung Cancer
Keywords: lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Arm (Experimental): Single Arm
  Interventions: Radiation: 4D-CT pre-treatment scan

INTERVENTIONS:
Radiation: 4D-CT pre-treatment scan — Undergo pre-treatment 4D-CT study for treatment planning External Beam Radiation: standard fractionation (2Gy per day) or stereotactic body radiation therapy Evaluation: Repeat 4D-CT study at 3 months and 6 months post-treatment
  Other Names: planning External Beam Radiation,; 4D-CT study

SUMMARY:
Eligible lung cancer patients: Undergo pre-treatment 4D-CT study for treatment planning

External Beam Radiation: standard fractionation (2Gy per day) or stereotactic body radiation therapy

Evaluation: Repeat 4D-CT study at 3 months and 6 months post-treatment

Primary objectives: To assess pre-treatment global and focal lung strain and correlate with changes post-treatment

DETAILED DESCRIPTION:
The study will be a prospective, non-randomized, single center, trial to assess and quantify lung strain using four dimensional CT (4D-CT) treatment planning scans. Patients with newly diagnosed lung cancer will be planned using 4D-CT to assess lung and tumor motion. Standard radiation treatment plans will to delivered based on tumor stage. Patients will be reassessed both clinically and radiographically using 4D-CT imaging at 3 months and 6 months post-treatment. Following the initial imaging time points, standard surveillance will be employed with clinical assessment and imaging at 3 month intervals for the first 2 years post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 18 years
2. ECOG performance status 0-1
3. Pathologic or clinical diagnosis of lung malignancy
4. Patients must have a reproducible tidal volume sufficient for 4D-CT imaging
5. Negative serum pregnancy test within 2 weeks prior to registration for women of childbearing potential.
6. Women of childbearing potential and male participants who are sexually active must agree to use a medically effective means of birth control
7. Patients must provide study specific informed consent prior to study entry.

Exclusion Criteria:

1. Patients with severe pulmonary dysfunction with non-reproducible tidal volumes sufficient for 4D-CT imaging.
2. Pregnant women or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-01; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
validate lung strain modeling using 4D-CT in a lung cancer patient population to correlate pre-treatment strain with post-treatment changes. | Pre-treatment (baseline) up to 6 months post-treatment
  The study will be a prospective, non-randomized, single center, trial to assess and quantify lung strain using 4D-CT treatment planning scans.

SECONDARY OUTCOMES:
correlate 4D-CT based lung strain modeling with standard lung function studies including pulmonary function tests and ventilation-perfusion scans. | 2 years post treatment
  4D-CT based lung strain modeling comparison with standard lung function
correlate pre- and post-treatment strain with clinical toxicity | Pre-treatment (baseline) to 2 years post treatment
  Toxicity correlation
correlate post-treatment strain with radiographic changes to the lung parenchyma | 2 years post-treatment
  Lung parenchyma correlation

CONTACTS AND LOCATIONS:
Overall Officials: Neal E Dunlap, MD, Principal Investigator — James Graham Brown Cancer Center
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States